CLINICAL TRIAL: NCT02921997
Title: A Phase II Study to Evaluate and Compare the Immunogenicity of Monovalent Inactivated Influenza A/H7N9 Virus Vaccine Administered With and Without AS03 Adjuvant and Monovalent Inactivated Influenza A/H3N2v Virus Vaccine Administered Without Adjuvant in Healthy Adults Through Standard and Systems Biology Analyses
Brief Title: H7N9 Vaccination With and Without AS03 and Unadjuvanted H3N2v Vaccination: Standard and Systems Biology Analyses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0015
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2019-08-08

CONDITIONS: Avian Influenza; H1N1 Influenza; Influenza
Keywords: A/H5N1; A/H7N9; ASO3 Adjuvant; influenza; monovalent; pH1N1; vaccines
MeSH Terms: conditions — Influenza in Birds; Orthomyxoviridae Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): 10 Subjects: one dose of 15 µg of A/H3N2v, at Day 1
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203
- Arm 2 (Experimental): 10 Subjects: two doses of 3.75 µg of AH7N9 AS03,at Day 1 and at Day 29
  Interventions: Drug: AS03; Biological: Monovalent influenza A/H7N9 virus vaccine
- Arm 3 (Experimental): 10 Subjects: two doses of 3.75 µg of A/H7N9, at Day 1 and Day 29
  Interventions: Biological: Monovalent influenza A/H7N9 virus vaccine

INTERVENTIONS:
Drug: AS03 — AS03 oil-in-water emulsion adjuvant.
  Arms: Arm 2
Biological: Influenza Virus Vaccine, Monovalent A/H3N2v A/Minnesota/11/2010 NYMC X-203 — Inactivated monovalent subvirion H3N2v vaccine containing hemagglutinin (HA) of A/Minnesota/11/2010 NYMC X-203 virus.
  Arms: Arm 1
Biological: Monovalent influenza A/H7N9 virus vaccine — Monovalent influenza A/H7N9 virus vaccine.
  Arms: Arm 2; Arm 3

SUMMARY:
This is a single center, randomized, partially-blinded, Phase II, small, targeted, prospective study in approximately 30 healthy male and non-pregnant female subjects aged 18 to 49 years old, inclusive, designed to evaluate and compare the immunogenicity between an intramuscular monovalent inactivated influenza A/H7N9 virus vaccine given with and without AS03 adjuvant, and an intramuscular unadjuvanted monovalent inactivated influenza A/H3N2v virus vaccine. The primary objectives are (1) assessing the serum anti-HA hemagglutination-inhibition (HAI) response to influenza A/H7N9 antigen (with and without adjuvant) at Day 57 (approximately one month after the second study vaccination with A/H7N9 vaccine with or without AS03) and influenza A/H3N2v antigen at Day 29 (approximately one month after the study vaccination with A/H3N2v), and (2) identifying differentially expressed genes in human immune cells on Days 2, 4, and 29 (following the first study vaccination with A/H7N9 vaccine with or without AS03) and on Days 30, 32, and 36 (following the second study vaccination with A/H7N9 vaccine with or without AS03), compared to baseline assessments performed prior to each study vaccination (Days -7, 1, and 29).

DETAILED DESCRIPTION:
This is a single center, randomized, partially-blinded, Phase II, small, targeted, prospective study in approximately 30 healthy male and non-pregnant female subjects aged 18 to 49 years old, inclusive, designed to evaluate and compare the immunogenicity between an intramuscular monovalent inactivated influenza A/H7N9 virus vaccine manufactured by Sanofi Pasteur given with and without AS03 adjuvant manufactured by GlaxoSmithKline, and an intramuscular unadjuvanted monovalent inactivated influenza A/H3N2v virus vaccine manufactured by Sanofi Pasteur. The primary objectives are (1) assessing the serum anti-HA hemagglutination-inhibition (HAI) response to influenza A/H7N9 antigen (with and without adjuvant) at Day 57 (approximately one month after the second study vaccination with A/H7N9 vaccine with or without AS03) and influenza A/H3N2v antigen at Day 29 (approximately one month after the study vaccination with A/H3N2v), and (2) identifying differentially expressed genes in human immune cells on Days 2, 4, and 29 (following the first study vaccination with A/H7N9 vaccine with or without AS03) and on Days 30, 32, and 36 (following the second study vaccination with A/H7N9 vaccine with or without AS03), compared to baseline assessments performed prior to each study vaccination (Days -7, 1, and 29). The secondary objectives are: (1) compare plasma cytokine and chemokine profiles at specific time points and between treatment arms at post vaccination points, (2) assess the neutralizing antibody responses to influenza A/H7N9 antigen (with and without adjuvant) at Day 57 (approximately one month after the second study vaccination with A/H7N9 vaccine with or without AS03) and influenza A/H3N2v antigen at Day 29 (approximately one month after the study vaccination with A/H3N2v vaccine), and (3) identify differentially expressed genes in human immune cells on Days 2, 4, and 8 following one intramuscular dose of influenza A/H3N2v vaccine compared to baseline assessments performed prior to study vaccination (Day -7 and Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 18 to 49 years old, inclusive.
4. Are in good health*.

   *As determined by medical history and targeted physical examination, if indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, that would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.4 degrees F.
6. Pulse is 50 to 115 bpm, inclusive.
7. Systolic blood pressure is 85 to 150 mm Hg, inclusive.
8. Diastolic blood pressure is 55 to 95 mm Hg, inclusive.
9. Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour.
10. Women of childbearing potential* must use an acceptable contraception method** from 30 days before first study vaccination until 60 days after last study vaccination.

    *Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

    **Includes, but is not limited to, non-male sexual relationships abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing (R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
11. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute or chronic medical disease or condition, defined as persisting for at least 90 days that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
4. Have known active neoplastic disease (excluding non-melanoma skin cancer) or a history of any hematologic malignancy.
5. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccines.
7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
8. Have a personal or family history of narcolepsy.
9. Have a history of Guillain-Barré syndrome.
10. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
11. Have a history of a potentially immune-mediated medical condition.
12. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
13. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
14. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
15. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
16. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as >840 mcg/day of beclomethasone dipropionate CFC or equivalent.
17. Received licensed live vaccine within 30 days prior to the first study vaccination, or plans to receive licensed live vaccine within 30 days before or after each study vaccination.
18. Received licensed inactivated vaccine within 14 days prior to the first study vaccination, or plans to receive licensed inactivated vaccine within 14 days before or after each study vaccination.
19. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
20. Received an experimental agent* within 30 days prior to the first study vaccination, or expects to receive an experimental agent** during the 13-month study-reporting period.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this study.
21. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the 13-month study-reporting period.

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
22. Prior participation in a clinical trial of influenza A/H7 vaccine* or have a history of influenza A/H7 virus actual or potential exposure or infection prior to the first study vaccination.

    *And assigned to a group receiving influenza A/H7 vaccine, does not apply to documented placebo recipients.
23. Prior participation in a clinical trial of influenza A/H3N2v vaccine* or have a history of influenza A/H3N2v virus actual or potential exposure or infection prior to the first study vaccination.

    *And assigned to a group receiving influenza A/H3N2v vaccine, does not apply to documented placebo recipients.
24. Occupational exposure to or substantial direct physical contact* with birds in the past year or during the 28 days after each study vaccination.

    *Casual contact with birds at petting zoos or county or state fairs or having pet birds does not exclude subjects from study participation.
25. Occupational exposure to or substantial direct physical contact* with pigs in the past year or during the 28 days after each study vaccination.

    *Casual contact with pigs at petting zoos or county or state fairs does not exclude subjects from study participation.
26. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
27. Plan to travel outside the US (continental US, Hawaii, and Alaska) within 28 days after each study vaccination.
28. Blood donation or planned blood donation within 30 days before enrollment until 30 days after the last blood draw for this study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center - Vanderbilt Institute for Clinical and Translational Research - Clinical Research Center (VICTR-CRC), Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females aged 18 to 49 years old, inclusively. They were recruited from the community at large around the clinic site. Participants were enrolled between 07NOV2016 and 31JAN2017.
Groups:
- A/H3N2v: One dose of 15 ug of A/H3N2v at Day 1
  A/H3N2v influenza virus vaccine: Monovalent inactivated influenza A/H3N2v virus vaccine (A/Minnesota/11/2010)
- A/H7N9 + AS03: Two doses of 3.75 ug of A/H7N9 + AS03, at Day 1 and Day 29 (+/- 2 days)
  AS03: AS03 oil-in-water emulsion adjuvant.
  A/H7N9 influenza virus vaccine: Monovalent inactivated influenza A/H7N9 virus vaccine (A/Shanghai/2/2013)
- A/H7N9: Two doses of 3.75 ug of A/H7N9, at Day 1 and Day 29 (+/- 2 days)
  A/H7N9 influenza virus vaccine: Monovalent inactivated influenza A/H7N9 virus vaccine (A/Shanghai/2/2013)
Period: Overall Study
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A/H3N2v: One dose of 15 ug of A/H3N2v, at Day 1 A/H3N2v influenza virus vaccine: Monovalent inactivated influenza A/H3N2v virus vaccine (A/Minnesota/11/2010).
- Total: Total of all reporting groups
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (7.1) | 28.0 (6.2) | 33.7 (8.3) | 30.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 5 | 19
  Male | 3 | 3 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.125 (5.609) | 21.885 (2.520) | 28.453 (10.768) | 24.821 (7.443)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroconversion Based on HAI Titer (A/H7N9 Vaccine, With and Without Adjuvant)
Description: Seroconversion is defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer =>1:40 or a pre-vaccination HAI titer =>1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer. Venous blood samples for serum were used for this assay. HAI based on the H7N9 strain A/Shanghai/02/2013xPR8 were assessed.
Time Frame: Day 29 Post-Vaccination 2 (Day 57)
Population: The intent-to-treat (ITT) population, A/H7N9 + AS03 and A/H7N9 arms: Includes all participants in the A/H7N9 + AS03 and A/H7N9 arms who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination blood samples for serological assessment (HAI or Neut antibody assays) for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- A/H7N9 + AS03: Two doses of 3.75 ug of monovalent inactivated influenza A/H7N9 virus vaccine with AS03 adjuvant at Day 1 and Day 29
- A/H7N9: Two doses of 3.75 ug of monovalent inactivated influenza A/H7N9 virus vaccine at Day 1 and Day 29
Arm/Group | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10
percentage of participants | 80.0 [44.4 to 97.5] | 0 [0.0 to 30.8]

2. Primary Outcome: Percentage of Participants Achieving Seroconversion Based on HAI Titer (A/H3N2v Vaccine)
Description: Seroconversion is defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer =>1:40 or a pre-vaccination HAI titer =>1:10 and a minimum four-fold rise in post-vaccination HAI antibody titer. Venous blood samples for serum were used for this assay. HAI based on the H3N2 strain A/Minnesota/11/2010 were assessed.
Time Frame: Day 29 Post-Vaccination 1 (Day 29)
Population: The intent-to-treat (ITT) population, A/H3N2v arm: Includes all participants in the A/H3N2v arm who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination blood samples for serological assessment (HAI or Neut antibody assays) for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- A/H3N2v: One dose of 15 ug monovalent inactivated influenza A/H3N2v virus vaccine at Day 1
Arm/Group | A/H3N2v
Number analyzed (Participants) | 10
percentage of participants | 50 [18.7 to 81.3]

3. Primary Outcome: Number of Differentially Expressed Genes Based on RNA Expression in Human Immune Cells (A/H7N9 Vaccine, With and Without Adjuvant)
Description: RNA expression levels (read counts) for each gene were determined by RNA-Sequencing of RNA extracted from six separated cell types: monocytes , dendritic cells, neutrophils, NK cells, B cells, and T cells. Post-vaccination gene expression levels were compared to pre-vaccination gene expression levels (combined summed read counts for Day -7 and Day 1 samples for post-vaccination 1 timepoints and Day 29 read counts for post-vaccination 2 timepoints) using a negative binomial model to identify differentially expressed (DE) genes (FDR-adjusted p-value < 0.05 and mean fold change => 1.5 in either direction).
Time Frame: Days 2, 4, and 29 Post-Vaccination 1 (Day 2, 4, and 29, respectively); Days 2, 4, and 8 Post-Vaccination 2 (Day 30, 32, and 36, respectively)
Population: The transcriptomics analysis population, A/H7N9 + AS03 and A/H7N9 arms: Includes all participants in the A/H7N9 +AS03 and A/H7N9 arms who received at least one study vaccination and contributed at least one pre- and one post-vaccination sample for transcriptomics testing for which valid results were reported.
Measure: Number; unit: Number of DE genes
Arm/Group | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10
Number of DE genes
  Monocytes : Day 2 Post Vaccination 1 | 618 | 0
  Monocytes : Day 4 Post Vaccination 1 | 36 | 0
  Monocytes : Day 29 Post Vaccination 1 | 0 | 0
  Monocytes : Day 2 Post Vaccination 2 | 1418 | 0
  Monocytes : Day 4 Post Vaccination 2 | 26 | 0
  Monocytes : Day 8 Post Vaccination 2 | 4 | 0
  Dendritic cells : Day 2 Post Vaccination 1 | 1091 | 0
  Dendritic cells : Day 4 Post Vaccination 1 | 8 | 0
  Dendritic cells : Day 29 Post Vaccination 1 | 1 | 0
  Dendritic cells : Day 2 Post Vaccination 2 | 1953 | 0
  Dendritic cells : Day 4 Post Vaccination 2 | 25 | 0
  Dendritic cells : Day 8 Post Vaccination 2 | 170 | 0
  Neutrophils : Day 2 Post Vaccination 1 | 1116 | 0
  Neutrophils : Day 4 Post Vaccination 1 | 41 | 0
  Neutrophils : Day 29 Post Vaccination 1 | 0 | 0
  Neutrophils : Day 2 Post Vaccination 2 | 2044 | 0
  Neutrophils : Day 4 Post Vaccination 2 | 181 | 0
  Neutrophils : Day 8 Post Vaccination 2 | 0 | 0
  NK cells : Day 2 Post Vaccination 1 | 60 | 0
  NK cells : Day 4 Post Vaccination 1 | 66 | 0
  NK cells : Day 29 Post Vaccination 1 | 8 | 0
  NK cells : Day 2 Post Vaccination 2 | 303 | 2
  NK cells : Day 4 Post Vaccination 2 | 396 | 0
  NK cells : Day 8 Post Vaccination 2 | 166 | 0
  B cells : Day 2 Post Vaccination 1 | 51 | 0
  B cells : Day 4 Post Vaccination 1 | 1 | 1
  B cells : Day 29 Post Vaccination 1 | 1 | 0
  B cells : Day 2 Post Vaccination 2 | 345 | 0
  B cells : Day 4 Post Vaccination 2 | 99 | 0
  B cells : Day 8 Post Vaccination 2 | 67 | 0
  T cells : Day 2 Post Vaccination 1 | 88 | 0
  T cells : Day 4 Post Vaccination 1 | 0 | 1
  T cells : Day 29 Post Vaccination 1 | 1 | 0
  T cells : Day 2 Post Vaccination 2 | 301 | 0
  T cells : Day 4 Post Vaccination 2 | 3 | 0
  T cells : Day 8 Post Vaccination 2 | 3 | 0

4. Secondary Outcome: Number of Differentially Expressed Genes Based on RNA Expression in Human Immune Cells (A/H3N2v Vaccine)
Description: RNA expression levels (read counts) for each gene were determined by RNA-Sequencing of RNA extracted from six separated cell types: monocytes, dendritic cells, neutrophils, NK cells, B cells, and T cells. Post-vaccination gene expression levels were compared to pre-vaccination gene expression levels (combined summed read counts for Day -7 and Day 1 samples for post-vaccination 1 timepoints) using a negative binomial model to identify differentially expressed (DE) genes (FDR-adjusted p-value < 0.05 and mean fold change => 1.5 in either direction).
Time Frame: Days 2, 4, and 8 Post-Vaccination 1 (Day 2, 4, and 8, respectively)
Population: The transcriptomics analysis population A/H3N2v arm: Includes all participants in the A/H3N2v arm who received at least one study vaccination and contributed at least one pre- and one post vaccination sample for transcriptomics testing for which valid results were reported.
Measure: Number; unit: Number of DE genes
Arm/Group | A/H3N2v
Number analyzed (Participants) | 10
Number of DE genes
  Monocytes : Day 2 Post Vaccination 1 | 0
  Monocytes : Day 4 Post Vaccination 1 | 0
  Monocytes : Day 8 Post Vaccination 1 | 1
  Dendritic cells : Day 2 Post Vaccination 1 | 0
  Dendritic cells : Day 4 Post Vaccination 1 | 0
  Dendritic cells : Day 8 Post Vaccination 1 | 2
  Neutrophils : Day 2 Post Vaccination 1 | 0
  Neutrophils : Day 4 Post Vaccination 1 | 0
  Neutrophils : Day 8 Post Vaccination 1 | 41
  NK cells : Day 2 Post Vaccination 1 | 0
  NK cells : Day 4 Post Vaccination 1 | 0
  NK cells : Day 8 Post Vaccination 1 | 1
  B cells : Day 2 Post Vaccination 1 | 0
  B cells : Day 4 Post Vaccination 1 | 0
  B cells : Day 8 Post Vaccination 1 | 3
  T cells : Day 2 Post Vaccination 1 | 0
  T cells : Day 4 Post Vaccination 1 | 0
  T cells : Day 8 Post Vaccination 1 | 0

5. Secondary Outcome: Cytokine and Chemokine Concentration by Study Arm and Study Visit Day - Part 1
Description: Venous blood samples for plasma were used for this assay. A Luminex assay was used to measure concentrations in ng/L. Concentrations for 11 of the total 24 cytokines and chemokines were measured: Fractalkine, Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF), Interferon-Gamma-Induced Protein-10(IP-10), Interferon-Alpha (IFNa), Interferon-Beta (IFNb), Interferon-Gamma (IFNy), Interferon-inducible T Cell Alpha Chemoattractant (ITAC), Interleukin 1 Beta (IL-1b), Interleukin 10 (IL-10), Interleukin 13 (IL-13), and Interleukin 2 (IL-2).
  If no cytokine or chemokine measurements were collected, number of participants is reported as 0.
Time Frame: Day 1 Pre-Vaccination 1; Days 2, 4, 8, and 29 Post-Vaccination 1 (Day 2, 4, 8, and 29, respectively); Days 2, 4, and 8 Post-Vaccination 2 (Day 30, 32, and 36, respectively)
Population: The intent-to-treat (ITT) population: Includes all participants who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination blood samples for serological assessment (HAI or Neut antibody assays) for which valid results were reported.
Measure: Median (95% Confidence Interval); unit: ng/L
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10 | 10
ng/L
  Fractalkine : Day 1 Pre-Vaccination | 310.9 [184.35 to 624.88] | 288.58 [177.74 to 489.88] | 356.19 [247.36 to 435.40]
  Fractalkine : Day 2 Post-Vaccination 1 | 312.26 [201.01 to 590.01] | 224.58 [181.26 to 530.97] | 315.31 [218.69 to 514.56]
  Fractalkine : Day 4 Post-Vaccination 1 | 345.14 [218.03 to 567.98] | 378.46 [172.26 to 543.87] | 309.48 [212.57 to 494.90]
  Fractalkine : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  Fractalkine : Day 8 Post-Vaccination 1 | 370.77 [204.33 to 783.22] |  |
  Fractalkine : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 29 Post-Vaccination 1 |  | 353.48 [210.90 to 492.30] | 333.38 [265.87 to 450.44]
  Fractalkine : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 2 Post-Vaccination 2 |  | 282.53 [178.94 to 566.01] | 305.83 [235.42 to 476.17]
  Fractalkine : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 4 Post-Vaccination 2 |  | 311.15 [223.31 to 466.89] | 316.25 [235.51 to 461.43]
  Fractalkine : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 8 Post-Vaccination 2 |  | 318.38 [178.94 to 486.64] | 306.53 [209.59 to 449.82]
  GM-CSF : Day 1 Pre-Vaccination | 511.59 [322.67 to 819.37] | 290.44 [188.18 to 447.68] | 478.50 [320.57 to 837.17]
  GM-CSF : Day 2 Post-Vaccination 1 | 557.77 [354.92 to 783.59] | 301.31 [195.59 to 423.36] | 478.66 [327.51 to 713.41]
  GM-CSF : Day 4 Post-Vaccination 1 | 561.63 [311.31 to 787.86] | 286.35 [171.87 to 477.21] | 448.62 [329.53 to 722.50]
  GM-CSF : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  GM-CSF : Day 8 Post-Vaccination 1 | 494.07 [238.89 to 778.82] |  |
  GM-CSF : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 29 Post-Vaccination 1 |  | 324.61 [192.61 to 392.17] | 476.40 [315.83 to 832.99]
  GM-CSF : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 2 Post-Vaccination 2 |  | 313.25 [225.34 to 442.63] | 497.90 [301.38 to 809.71]
  GM-CSF : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 4 Post-Vaccination 2 |  | 259.34 [210.99 to 385.57] | 468.16 [344.33 to 920.82]
  GM-CSF : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 8 Post-Vaccination 2 |  | 276.04 [195.20 to 452.95] | 468.95 [330.08 to 612.07]
  IP-10 : Day 1 Pre-Vaccination | 249.16 [209.78 to 360.45] | 288.09 [194.27 to 444.35] | 238.80 [157.18 to 324.89]
  IP-10 : Day 2 Post-Vaccination 1 | 261.78 [229.52 to 621.71] | 535.80 [372.78 to 709.82] | 273.48 [137.01 to 362.69]
  IP-10 : Day 4 Post-Vaccination 1 | 242.77 [198.72 to 376.06] | 417.82 [263.11 to 560.03] | 219.79 [161.22 to 381.36]
  IP-10 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IP-10 : Day 8 Post-Vaccination 1 | 236.95 [175.75 to 315.67] |  |
  IP-10 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 29 Post-Vaccination 1 |  | 284.62 [200.09 to 367.84] | 212.26 [144.78 to 259.60]
  IP-10 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 2 Post-Vaccination 2 |  | 1264.00 [586.12 to 2541.12] | 234.75 [134.66 to 311.02]
  IP-10 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 4 Post-Vaccination 2 |  | 512.16 [339.91 to 567.27] | 224.40 [154.65 to 322.71]
  IP-10 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 8 Post-Vaccination 2 |  | 307.23 [227.78 to 373.61] | 220.60 [127.68 to 280.31]
  IFNa : Day 1 Pre-Vaccination | 116.80 [58.27 to 149.96] | 142.43 [91.50 to 213.19] | 104.81 [64.58 to 152.56]
  IFNa : Day 2 Post-Vaccination 1 | 73.98 [62.82 to 155.25] | 132.03 [91.88 to 179.71] | 101.40 [38.58 to 232.97]
  IFNa : Day 4 Post-Vaccination 1 | 66.93 [30.39 to 191.17] | 125.29 [87.21 to 251.48] | 86.82 [29.60 to 181.88]
  IFNa : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNa : Day 8 Post-Vaccination 1 | 89.29 [51.11 to 153.41] |  |
  IFNa : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 29 Post-Vaccination 1 |  | 118.90 [79.39 to 218.86] | 111.00 [53.91 to 149.95]
  IFNa : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 2 Post-Vaccination 2 |  | 130.25 [97.22 to 213.06] | 89.99 [38.72 to 161.13]
  IFNa : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 4 Post-Vaccination 2 |  | 127.23 [93.43 to 231.92] | 113.26 [51.80 to 225.69]
  IFNa : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 8 Post-Vaccination 2 |  | 163.86 [102.50 to 219.70] | 89.00 [26.83 to 168.33]
  IFNb : Day 1 Pre-Vaccination | 1073.70 [856.91 to 1843.25] | 1211.25 [743.26 to 1686.50] | 989.57 [760.70 to 1818.92]
  IFNb : Day 2 Post-Vaccination 1 | 1023.11 [732.33 to 1286.00] | 1068.38 [708.26 to 1620.50] | 1106.50 [657.21 to 1516.84]
  IFNb : Day 4 Post-Vaccination 1 | 878.76 [735.36 to 1534.50] | 1074.52 [739.07 to 1730.00] | 1045.50 [867.77 to 1768.00]
  IFNb : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNb : Day 8 Post-Vaccination 1 | 1104.00 [718.50 to 1564.00] |  |
  IFNb : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 29 Post-Vaccination 1 |  | 1185.00 [598.46 to 1407.50] | 1109.00 [684.26 to 2134.00]
  IFNb : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 2 Post-Vaccination 2 |  | 1188.50 [734.74 to 1757.00] | 1241.50 [624.16 to 1883.74]
  IFNb : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 4 Post-Vaccination 2 |  | 1027.74 [649.67 to 1760.00] | 980.99 [776.21 to 1564.00]
  IFNb : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 8 Post-Vaccination 2 |  | 992.82 [647.85 to 1671.50] | 1326.50 [776.40 to 1521.25]
  IFNy : Day 1 Pre-Vaccination | 28.71 [13.21 to 46.65] | 17.86 [11.28 to 43.92] | 33.82 [22.85 to 45.92]
  IFNy : Day 2 Post-Vaccination 1 | 26.47 [12.49 to 54.72] | 21.22 [13.01 to 47.81] | 33.17 [22.11 to 46.45]
  IFNy : Day 4 Post-Vaccination 1 | 26.38 [14.20 to 50.92] | 19.01 [9.02 to 47.74] | 33.74 [22.81 to 41.58]
  IFNy : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNy : Day 8 Post-Vaccination 1 | 30.98 [13.45 to 48.70] |  |
  IFNy : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 29 Post-Vaccination 1 |  | 23.07 [11.57 to 49.17] | 32.43 [25.74 to 39.04]
  IFNy : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 2 Post-Vaccination 2 |  | 37.22 [23.07 to 59.78] | 30.79 [25.01 to 36.40]
  IFNy : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 4 Post-Vaccination 2 |  | 19.99 [10.90 to 41.65] | 29.70 [22.16 to 39.11]
  IFNy : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 8 Post-Vaccination 2 |  | 18.00 [11.37 to 46.89] | 28.94 [21.79 to 36.99]
  ITAC : Day 1 Pre-Vaccination | 58.19 [27.49 to 140.69] | 44.19 [30.64 to 76.83] | 52.62 [26.89 to 89.05]
  ITAC : Day 2 Post-Vaccination 1 | 56.31 [27.66 to 152.10] | 52.46 [35.90 to 90.02] | 49.22 [30.06 to 75.22]
  ITAC : Day 4 Post-Vaccination 1 | 51.68 [23.65 to 188.54] | 47.38 [36.63 to 84.94] | 52.83 [24.25 to 69.46]
  ITAC : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  ITAC : Day 8 Post-Vaccination 1 | 49.21 [20.12 to 205.30] |  |
  ITAC : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 29 Post-Vaccination 1 |  | 60.62 [23.95 to 86.14] | 49.58 [24.37 to 68.83]
  ITAC : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 2 Post-Vaccination 2 |  | 77.16 [48.46 to 191.11] | 45.04 [23.91 to 68.24]
  ITAC : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 4 Post-Vaccination 2 |  | 58.32 [31.86 to 83.67] | 34.97 [24.36 to 59.44]
  ITAC : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 8 Post-Vaccination 2 |  | 50.94 [36.37 to 84.45] | 47.67 [28.41 to 76.88]
  IL-1b : Day 1 Pre-Vaccination | 2.84 [1.75 to 4.74] | 2.83 [1.43 to 5.08] | 3.33 [2.10 to 6.93]
  IL-1b : Day 2 Post-Vaccination 1 | 2.62 [1.68 to 4.57] | 2.33 [1.30 to 5.28] | 3.46 [2.22 to 7.00]
  IL-1b : Day 4 Post-Vaccination 1 | 2.78 [1.81 to 4.46] | 3.46 [1.34 to 5.80] | 3.39 [2.08 to 5.58]
  IL-1b : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-1b : Day 8 Post-Vaccination 1 | 2.82 [1.78 to 5.41] |  |
  IL-1b : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 29 Post-Vaccination 1 |  | 3.25 [1.67 to 5.49] | 3.70 [2.25 to 5.03]
  IL-1b : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 2 Post-Vaccination 2 |  | 2.99 [1.37 to 7.12] | 3.88 [2.12 to 5.63]
  IL-1b : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 4 Post-Vaccination 2 |  | 2.81 [1.49 to 4.93] | 3.16 [2.25 to 6.93]
  IL-1b : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 8 Post-Vaccination 2 |  | 2.52 [1.59 to 7.03] | 3.03 [2.15 to 5.20]
  IL-10 : Day 1 Pre-Vaccination | 21.92 [9.32 to 59.45] | 18.28 [10.29 to 37.48] | 27.67 [19.96 to 40.21]
  IL-10 : Day 2 Post-Vaccination 1 | 22.26 [10.43 to 65.61] | 17.16 [13.04 to 38.18] | 26.04 [21.00 to 36.63]
  IL-10 : Day 4 Post-Vaccination 1 | 22.29 [15.03 to 72.99] | 17.64 [12.84 to 39.04] | 29.53 [20.68 to 41.65]
  IL-10 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-10 : Day 8 Post-Vaccination 1 | 19.52 [12.57 to 105.24] |  |
  IL-10 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 29 Post-Vaccination 1 |  | 19.93 [12.35 to 38.28] | 26.71 [21.28 to 36.63]
  IL-10 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 2 Post-Vaccination 2 |  | 23.79 [11.07 to 44.81] | 24.57 [17.44 to 35.06]
  IL-10 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 4 Post-Vaccination 2 |  | 19.29 [14.95 to 36.55] | 26.39 [17.73 to 38.52]
  IL-10 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 8 Post-Vaccination 2 |  | 21.75 [12.06 to 35.99] | 23.29 [19.25 to 31.83]
  IL-13 : Day 1 Pre-Vaccination | 11.24 [6.18 to 33.79] | 18.39 [8.41 to 28.27] | 12.46 [8.35 to 21.16]
  IL-13 : Day 2 Post-Vaccination 1 | 10.98 [6.97 to 39.49] | 20.66 [8.93 to 25.85] | 11.72 [8.01 to 23.73]
  IL-13 : Day 4 Post-Vaccination 1 | 13.86 [6.33 to 39.49] | 21.10 [9.03 to 25.98] | 11.51 [7.94 to 22.80]
  IL-13 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-13 : Day 8 Post-Vaccination 1 | 11.02 [5.48 to 61.06] |  |
  IL-13 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 29 Post-Vaccination 1 |  | 19.35 [10.85 to 33.12] | 10.80 [5.79 to 21.52]
  IL-13 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 2 Post-Vaccination 2 |  | 18.99 [9.84 to 36.55] | 10.79 [6.40 to 20.43]
  IL-13 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 4 Post-Vaccination 2 |  | 17.56 [11.01 to 35.15] | 10.08 [6.55 to 20.46]
  IL-13 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 8 Post-Vaccination 2 |  | 21.50 [8.16 to 39.16] | 10.36 [7.25 to 21.45]
  IL-2 : Day 1 Pre-Vaccination | 3.30 [2.02 to 6.67] | 2.49 [1.33 to 6.58] | 4.48 [2.73 to 8.18]
  IL-2 : Day 2 Post-Vaccination 1 | 4.13 [1.94 to 6.52] | 2.52 [1.20 to 6.57] | 4.32 [2.77 to 8.76]
  IL-2 : Day 4 Post-Vaccination 1 | 3.43 [2.03 to 6.49] | 2.28 [1.74 to 7.00] | 3.82 [2.98 to 7.79]
  IL-2 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-2 : Day 8 Post-Vaccination 1 | 2.99 [2.62 to 7.74] |  |
  IL-2 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 29 Post-Vaccination 1 |  | 2.29 [1.77 to 7.40] | 4.68 [3.08 to 6.97]
  IL-2 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 2 Post-Vaccination 2 |  | 2.39 [1.17 to 8.47] | 4.05 [2.64 to 8.21]
  IL-2 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 4 Post-Vaccination 2 |  | 2.71 [1.46 to 6.85] | 3.74 [2.69 to 9.81]
  IL-2 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 8 Post-Vaccination 2 |  | 3.14 [1.70 to 6.84] | 3.97 [2.69 to 6.22]

6. Secondary Outcome: Cytokine and Chemokine Concentration by Study Arm and Study Visit Day - Part 2
Description: Venous blood samples for plasma were used for this assay. A Luminex assay was used to measure concentrations in ng/L. Concentrations for 9 of the total 24 cytokines and chemokines were measured: Interleukin 21 (IL-21), Interleukin 23 (IL-23), Interleukin 4 (IL-4), Interleukin 5 (IL-5), Interleukin 6 (IL-6), Interleukin 7 (IL-7), Interleukin 8 (IL-8), Interleukin 12, p70 (IL-12p70), and Interleukin 17A (IL-17A).
  If no cytokine or chemokine measurements were collected, number of participants is reported as 0.
Time Frame: as for outcome 5
Population: The intent-to-treat (ITT) population: Includes all participants who received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination blood samples for serological assessment (HAI or Neut antibody assays) for which valid results were reported. No cytokine or chemokine measurements were collected for the A/H3N2v arm after Day 8 Post-Vaccination 1 (Day 8), and for the A/H7N9 + AS03 and A/H7N9 arms at Day 8 Post-Vaccination 1 (Day 8).
Measure: Median (95% Confidence Interval); unit: ng/L
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10 | 10
ng/L
  IL-21 : Day 1 Pre-Vaccination | 3.54 [1.39 to 9.12] | 3.25 [1.64 to 4.33] | 2.43 [1.66 to 10.32]
  IL-21 : Day 2 Post-Vaccination 1 | 3.83 [1.56 to 10.25] | 3.00 [1.76 to 5.34] | 2.63 [1.76 to 9.32]
  IL-21 : Day 4 Post-Vaccination 1 | 4.47 [1.92 to 11.57] | 2.76 [1.90 to 5.22] | 2.64 [1.76 to 9.26]
  IL-21 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-21 : Day 8 Post-Vaccination 1 | 2.76 [1.12 to 15.81] |  |
  IL-21 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 29 Post-Vaccination 1 |  | 4.76 [1.90 to 5.77] | 2.53 [1.73 to 9.57]
  IL-21 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 2 Post-Vaccination 2 |  | 4.29 [2.13 to 6.54] | 2.09 [1.38 to 9.30]
  IL-21 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 4 Post-Vaccination 2 |  | 3.96 [1.96 to 5.91] | 2.01 [1.59 to 10.27]
  IL-21 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 8 Post-Vaccination 2 |  | 2.85 [1.84 to 6.78] | 1.93 [1.71 to 7.32]
  IL-23 : Day 1 Pre-Vaccination | 367.05 [245.03 to 565.32] | 368.23 [280.19 to 527.92] | 550.19 [340.63 to 750.07]
  IL-23 : Day 2 Post-Vaccination 1 | 304.56 [213.42 to 482.68] | 362.33 [199.20 to 495.74] | 490.16 [336.64 to 807.72]
  IL-23 : Day 4 Post-Vaccination 1 | 419.28 [222.30 to 569.42] | 468.30 [246.74 to 605.22] | 583.59 [328.03 to 786.52]
  IL-23 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-23 : Day 8 Post-Vaccination 1 | 339.06 [256.69 to 555.18] |  |
  IL-23 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 29 Post-Vaccination 1 |  | 418.57 [311.36 to 548.07] | 496.08 [317.22 to 918.63]
  IL-23 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 2 Post-Vaccination 2 |  | 487.09 [312.55 to 758.84] | 536.87 [345.26 to 768.30]
  IL-23 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 4 Post-Vaccination 2 |  | 409.82 [319.81 to 524.89] | 514.30 [310.06 to 768.41]
  IL-23 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 8 Post-Vaccination 2 |  | 421.69 [326.56 to 622.45] | 444.43 [341.61 to 916.35]
  IL-4 : Day 1 Pre-Vaccination | 61.67 [48.37 to 103.08] | 49.85 [39.70 to 119.83] | 59.30 [46.83 to 154.39]
  IL-4 : Day 2 Post-Vaccination 1 | 69.57 [43.44 to 105.29] | 53.00 [36.30 to 123.64] | 63.35 [45.19 to 188.85]
  IL-4 : Day 4 Post-Vaccination 1 | 68.54 [50.44 to 91.18] | 53.75 [37.06 to 128.56] | 58.21 [41.52 to 150.14]
  IL-4 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-4 : Day 8 Post-Vaccination 1 | 63.89 [41.87 to 106.36] |  |
  IL-4 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 29 Post-Vaccination 1 |  | 59.46 [42.24 to 132.19] | 59.83 [41.62 to 158.67]
  IL-4 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 2 Post-Vaccination 2 |  | 66.66 [33.95 to 135.48] | 61.47 [38.94 to 136.29]
  IL-4 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 4 Post-Vaccination 2 |  | 67.74 [35.01 to 121.38] | 59.86 [40.82 to 167.25]
  IL-4 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 8 Post-Vaccination 2 |  | 54.44 [39.43 to 159.90] | 63.96 [37.41 to 122.34]
  IL-5 : Day 1 Pre-Vaccination | 3.22 [1.54 to 6.26] | 3.92 [2.46 to 5.98] | 2.82 [2.16 to 7.27]
  IL-5 : Day 2 Post-Vaccination 1 | 3.04 [1.55 to 7.85] | 4.54 [2.46 to 5.53] | 2.84 [2.12 to 6.93]
  IL-5 : Day 4 Post-Vaccination 1 | 2.96 [1.45 to 7.93] | 4.73 [2.90 to 6.04] | 3.03 [1.79 to 8.55]
  IL-5 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-5 : Day 8 Post-Vaccination 1 | 2.50 [1.66 to 9.71] |  |
  IL-5 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 29 Post-Vaccination 1 |  | 4.56 [2.35 to 7.50] | 3.33 [2.08 to 6.96]
  IL-5 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 2 Post-Vaccination 2 |  | 4.83 [2.75 to 9.01] | 3.03 [1.88 to 6.98]
  IL-5 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 4 Post-Vaccination 2 |  | 4.15 [2.56 to 7.36] | 3.04 [2.17 to 7.92]
  IL-5 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 8 Post-Vaccination 2 |  | 4.78 [2.63 to 7.19] | 3.25 [1.77 to 6.43]
  IL-6 : Day 1 Pre-Vaccination | 2.02 [1.19 to 4.09] | 1.26 [0.86 to 5.33] | 3.39 [2.15 to 5.62]
  IL-6 : Day 2 Post-Vaccination 1 | 2.03 [1.30 to 5.00] | 2.54 [1.73 to 6.08] | 3.23 [2.17 to 6.54]
  IL-6 : Day 4 Post-Vaccination 1 | 2.09 [1.21 to 5.42] | 1.48 [0.72 to 4.23] | 3.39 [2.25 to 6.85]
  IL-6 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-6 : Day 8 Post-Vaccination 1 | 2.28 [0.75 to 4.52] |  |
  IL-6 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 29 Post-Vaccination 1 |  | 1.75 [0.98 to 3.60] | 3.52 [2.33 to 4.60]
  IL-6 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 2 Post-Vaccination 2 |  | 2.95 [2.20 to 4.60] | 3.09 [2.22 to 4.95]
  IL-6 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 4 Post-Vaccination 2 |  | 1.48 [0.99 to 3.31] | 3.06 [2.21 to 4.92]
  IL-6 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 8 Post-Vaccination 2 |  | 1.07 [0.71 to 3.33] | 3.11 [1.80 to 4.28]
  IL-7 : Day 1 Pre-Vaccination | 4.02 [2.50 to 8.88] | 4.58 [2.27 to 10.37] | 5.22 [3.62 to 10.88]
  IL-7 : Day 2 Post-Vaccination 1 | 3.90 [2.72 to 9.67] | 4.05 [1.75 to 11.04] | 5.12 [4.00 to 10.56]
  IL-7 : Day 4 Post-Vaccination 1 | 3.71 [2.35 to 6.81] | 4.93 [1.75 to 11.18] | 4.97 [3.37 to 12.30]
  IL-7 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-7 : Day 8 Post-Vaccination 1 | 3.89 [3.00 to 14.78] |  |
  IL-7 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 29 Post-Vaccination 1 |  | 5.85 [2.19 to 10.39] | 4.99 [4.06 to 9.92]
  IL-7 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 2 Post-Vaccination 2 |  | 6.20 [2.27 to 11.20] | 4.41 [3.44 to 9.50]
  IL-7 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 4 Post-Vaccination 2 |  | 5.56 [1.76 to 9.02] | 4.83 [3.04 to 9.12]
  IL-7 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 8 Post-Vaccination 2 |  | 5.46 [2.66 to 12.88] | 4.03 [3.13 to 9.96]
  IL-8 : Day 1 Pre-Vaccination | 4.37 [3.27 to 28.92] | 6.97 [3.31 to 9.79] | 5.53 [3.26 to 10.62]
  IL-8 : Day 2 Post-Vaccination 1 | 5.04 [4.03 to 16.04] | 6.76 [3.32 to 9.22] | 5.04 [3.14 to 10.18]
  IL-8 : Day 4 Post-Vaccination 1 | 4.86 [3.80 to 16.79] | 7.47 [3.11 to 10.11] | 5.33 [3.58 to 9.75]
  IL-8 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-8 : Day 8 Post-Vaccination 1 | 4.35 [3.50 to 24.83] |  |
  IL-8 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 29 Post-Vaccination 1 |  | 7.42 [2.90 to 9.27] | 4.53 [3.29 to 9.51]
  IL-8 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 2 Post-Vaccination 2 |  | 8.41 [2.73 to 12.62] | 4.84 [3.16 to 8.89]
  IL-8 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 4 Post-Vaccination 2 |  | 7.03 [2.11 to 10.18] | 4.70 [2.93 to 8.43]
  IL-8 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 8 Post-Vaccination 2 |  | 5.64 [2.98 to 11.70] | 4.44 [3.06 to 9.07]
  IL-12p70 : Day 1 Pre-Vaccination | 3.96 [1.67 to 7.55] | 2.53 [1.36 to 6.09] | 5.33 [1.82 to 9.53]
  IL-12p70 : Day 2 Post-Vaccination 1 | 3.93 [2.04 to 7.59] | 2.50 [1.40 to 6.32] | 4.18 [1.48 to 11.06]
  IL-12p70 : Day 4 Post-Vaccination 1 | 3.95 [1.88 to 7.66] | 2.68 [1.70 to 6.27] | 4.90 [2.05 to 9.85]
  IL-12p70 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-12p70 : Day 8 Post-Vaccination 1 | 4.63 [1.81 to 8.22] |  |
  IL-12p70 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 29 Post-Vaccination 1 |  | 3.65 [1.46 to 6.80] | 5.63 [1.64 to 7.53]
  IL-12p70 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 2 Post-Vaccination 2 |  | 3.83 [1.34 to 8.87] | 5.01 [1.84 to 7.65]
  IL-12p70 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 4 Post-Vaccination 2 |  | 3.69 [1.74 to 5.58] | 4.44 [2.33 to 8.64]
  IL-12p70 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 8 Post-Vaccination 2 |  | 2.18 [1.66 to 7.71] | 5.08 [1.67 to 8.29]
  IL-17A: Day 1 Pre-Vaccination | 19.44 [11.52 to 26.02] | 14.04 [9.60 to 33.02] | 24.34 [18.45 to 39.84]
  IL-17A : Day 2 Post-Vaccination 1 | 18.06 [11.27 to 29.38] | 15.12 [8.00 to 36.45] | 20.96 [16.61 to 38.07]
  IL-17A : Day 4 Post-Vaccination 1 | 20.03 [11.40 to 34.12] | 14.86 [9.26 to 35.99] | 22.84 [16.82 to 34.56]
  IL-17A : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-17A : Day 8 Post-Vaccination 1 | 22.21 [11.47 to 33.23] |  |
  IL-17A : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 29 Post-Vaccination 1 |  | 17.44 [9.81 to 37.00] | 23.83 [20.33 to 30.67]
  IL-17A : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 2 Post-Vaccination 2 |  | 18.69 [8.98 to 35.80] | 23.50 [18.52 to 30.20]
  IL-17A : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 4 Post-Vaccination 2 |  | 16.66 [9.39 to 32.65] | 21.67 [18.70 to 34.83]
  IL-17A : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 8 Post-Vaccination 2 |  | 13.24 [10.13 to 27.27] | 21.34 [16.22 to 30.88]

7. Secondary Outcome: Cytokine and Chemokine Concentration by Study Arm and Study Visit Day - Part 3
Description: Venous blood samples for plasma were used for this assay. A Luminex assay was used to measure concentrations in ng/L. Concentrations for 4 of the total 24 cytokines and chemokines were measured: Macrophage Inflammatory Protein-1 Alpha (MIP1a), Macrophage Inflammatory Protein-1 Beta (MIP1b), Macrophage Inflammatory Protein-3 Alpha (MIP3a), and Tumor Necrosis Factor Alpha (TNF-a).
  If no cytokine or chemokine measurements were collected, number of participants is reported as 0.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: ng/L
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10 | 10
ng/L
  MIP1a : Day 1 Pre-Vaccination | 25.49 [15.16 to 42.51] | 24.86 [17.98 to 38.64] | 22.98 [18.00 to 41.08]
  MIP1a : Day 2 Post-Vaccination 1 | 24.56 [14.79 to 43.50] | 24.96 [17.78 to 40.41] | 23.13 [16.62 to 45.80]
  MIP1a : Day 4 Post-Vaccination 1 | 23.86 [15.07 to 50.72] | 24.44 [19.50 to 37.41] | 22.34 [18.16 to 46.99]
  MIP1a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP1a : Day 8 Post-Vaccination 1 | 27.64 [16.04 to 54.73] |  |
  MIP1a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 29 Post-Vaccination 1 |  | 26.08 [18.52 to 36.89] | 23.09 [17.91 to 43.35]
  MIP1a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 2 Post-Vaccination 2 |  | 29.90 [22.66 to 39.17] | 21.25 [18.28 to 43.92]
  MIP1a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 4 Post-Vaccination 2 |  | 24.08 [17.70 to 38.31] | 23.44 [17.45 to 44.09]
  MIP1a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 8 Post-Vaccination 2 |  | 33.32 [15.40 to 41.68] | 22.54 [15.73 to 42.55]
  MIP1b : Day 1 Pre-Vaccination | 18.63 [15.69 to 31.89] | 12.99 [10.99 to 27.31] | 20.33 [14.53 to 36.98]
  MIP1b : Day 2 Post-Vaccination 1 | 20.43 [17.90 to 31.63] | 16.90 [12.06 to 33.56] | 19.84 [13.91 to 34.72]
  MIP1b : Day 4 Post-Vaccination 1 | 20.47 [16.69 to 27.61] | 14.76 [10.77 to 33.98] | 19.16 [15.58 to 40.36]
  MIP1b : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP1b : Day 8 Post-Vaccination 1 | 23.67 [16.79 to 37.81] |  |
  MIP1b : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 29 Post-Vaccination 1 |  | 16.05 [9.66 to 28.29] | 18.35 [12.76 to 35.12]
  MIP1b : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 2 Post-Vaccination 2 |  | 29.05 [18.38 to 40.59] | 16.78 [13.36 to 32.55]
  MIP1b : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 4 Post-Vaccination 2 |  | 14.42 [10.92 to 23.29] | 17.56 [14.29 to 36.42]
  MIP1b : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 8 Post-Vaccination 2 |  | 16.18 [10.86 to 28.51] | 16.18 [14.61 to 32.97]
  MIP3a : Day 1 Pre-Vaccination | 16.77 [11.10 to 32.16] | 15.34 [9.87 to 29.55] | 16.60 [12.26 to 33.44]
  MIP3a : Day 2 Post-Vaccination 1 | 19.59 [11.39 to 24.35] | 13.90 [8.92 to 25.28] | 15.44 [13.38 to 32.35]
  MIP3a : Day 4 Post-Vaccination 1 | 18.58 [10.93 to 27.55] | 16.49 [8.94 to 24.60] | 15.74 [14.29 to 29.96]
  MIP3a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP3a : Day 8 Post-Vaccination 1 | 18.62 [13.23 to 34.32] |  |
  MIP3a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 29 Post-Vaccination 1 |  | 15.72 [11.19 to 27.29] | 16.05 [12.70 to 34.47]
  MIP3a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 2 Post-Vaccination 2 |  | 16.24 [11.39 to 25.25] | 14.27 [11.30 to 31.88]
  MIP3a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 4 Post-Vaccination 2 |  | 16.24 [10.71 to 22.28] | 15.31 [12.46 to 40.70]
  MIP3a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 8 Post-Vaccination 2 |  | 19.01 [10.22 to 28.61] | 14.53 [12.18 to 50.55]
  TNF-a : Day 1 Pre-Vaccination | 4.32 [3.64 to 8.29] | 4.18 [2.66 to 7.11] | 5.36 [3.85 to 9.95]
  TNF-a : Day 2 Post-Vaccination 1 | 5.13 [3.75 to 8.30] | 4.26 [3.18 to 8.59] | 5.40 [3.32 to 10.16]
  TNF-a : Day 4 Post-Vaccination 1 | 5.16 [4.02 to 7.83] | 4.78 [3.21 to 9.07] | 5.24 [4.09 to 12.87]
  TNF-a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  TNF-a : Day 8 Post-Vaccination 1 | 4.48 [3.52 to 9.02] |  |
  TNF-a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 29 Post-Vaccination 1 |  | 4.88 [2.95 to 8.00] | 4.93 [3.20 to 10.11]
  TNF-a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 2 Post-Vaccination 2 |  | 8.13 [5.61 to 11.90] | 4.78 [3.19 to 9.54]
  TNF-a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 4 Post-Vaccination 2 |  | 5.28 [3.34 to 7.34] | 5.26 [3.03 to 11.05]
  TNF-a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 8 Post-Vaccination 2 |  | 4.56 [3.85 to 7.69] | 4.54 [3.23 to 9.62]

8. Secondary Outcome: Fold Change in Cytokine and Chemokine Concentrations From Pre-vaccination - Part 1
Description: Venous blood samples for plasma were used for this assay. A Luminex assay was used to measure concentrations in ng/L. Concentrations for 7 of the total 24 cytokines and chemokines were measured: Fractalkine, GM-CSF, IP-10, IFNa, IFNb, IFNy, and ITAC.
  If no cytokine or chemokine measurements were collected, number of participants is reported as 0.
Time Frame: Days 2, 4, 8, and 29 Post-Vaccination 1 (Day 2, 4, 8, and 29, respectively); Days 2, 4, and 8 Post-Vaccination 2 (Day 30, 32, and 36, respectively)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10 | 10
fold change
  Fractalkine : Day 2 Post-Vaccination 1 | 0.944 [0.850 to 1.170] | 1.015 [0.830 to 1.080] | 1.003 [0.870 to 1.070]
  Fractalkine : Day 4 Post-Vaccination 1 | 1.024 [0.910 to 1.350] | 1.092 [0.890 to 1.470] | 0.946 [.840 to 1.140]
  Fractalkine : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  Fractalkine : Day 8 Post-Vaccination 1 | 0.983 [0.920 to 1.160] |  |
  Fractalkine : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 29 Post-Vaccination 1 |  | 0.999 [0.900 to 1.240] | 1.063 [0.860 to 1.080]
  Fractalkine : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 2 Post-Vaccination 2 |  | 1.010 [0.860 to 1.300] | 1.053 [0.880 to 1.100]
  Fractalkine : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 4 Post-Vaccination 2 |  | 1.022 [0.800 to 1.130] | 1.010 [0.840 to 1.290]
  Fractalkine : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  Fractalkine : Day 8 Post-Vaccination 2 |  | 0.931 [.770 to 1.250] | 0.985 [0.880 to 1.100]
  GM-CSF : Day 2 Post-Vaccination 1 | 1.117 [1.00 to 1.220] | 1.020 [0.890 to 1.070] | 0.971 [0.920 to 1.090]
  GM-CSF : Day 4 Post-Vaccination 1 | 1.096 [0.960 to 1.200] | 0.932 [0.850 to 1.170] | 0.971 [0.860 to 1.100]
  GM-CSF : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  GM-CSF : Day 8 Post-Vaccination 1 | 1.043 [0.970 to 1.200] |  |
  GM-CSF : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 29 Post-Vaccination 1 |  | 1.053 [0.860 to 1.280] | 1.018 [0.960 to 1.070]
  GM-CSF : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 2 Post-Vaccination 2 |  | 1.107 [0.940 to 1.210] | 0.994 [0.900 to 1.060]
  GM-CSF : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 4 Post-Vaccination 2 |  | 0.832 [0.770 to 1.040] | 1.004 [0.900 to 1.170]
  GM-CSF : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  GM-CSF : Day 8 Post-Vaccination 2 |  | 1.053 [0.770 to 1.210] | 0.969 [0.900 to 1.010]
  IP-10 : Day 2 Post-Vaccination 1 | 0.988 [0.870 to 1.250] | 1.867 [0.990 to 2.740] | 1.065 [0.910 to 1.190]
  IP-10 : Day 4 Post-Vaccination 1 | 0.983 [0.760 to 1.090] | 1.445 [0.750 to 1.810] | 0.977 [0.850 to 1.150]
  IP-10 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IP-10 : Day 8 Post-Vaccination 1 | 0.889 [0.650 to 0.960] |  |
  IP-10 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 29 Post-Vaccination 1 |  | 0.869 [0.720 to 1.140] | 0.868 [0.780 to 0.930]
  IP-10 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 2 Post-Vaccination 2 |  | 4.461 [2.190 to 8.260] | 1.097 [1.030 to 1.340]
  IP-10 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 4 Post-Vaccination 2 |  | 1.450 [1.160 to 1.930] | 1.111 [0.970 to 1.340]
  IP-10 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IP-10 : Day 8 Post-Vaccination 2 |  | 1.002 [0.850 to 1.060] | 1.022 [0.910 to 1.250]
  IFNa : Day 2 Post-Vaccination 1 | 0.830 [0.620 to 1.090] | 0.959 [0.790 to 1.130] | 1.207 [0.600 to 2.040]
  IFNa : Day 4 Post-Vaccination 1 | 0.807 [0.380 to 1.250] | 1.023 [0.840 to 1.270] | 1.121 [0.470 to 1.270]
  IFNa : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNa : Day 8 Post-Vaccination 1 | 0.877 [0.550 to 1.300] |  |
  IFNa : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 29 Post-Vaccination 1 |  | 0.969 [0.640 to 1.260] | 0.924 [0.700 to 0.980]
  IFNa : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 2 Post-Vaccination 2 |  | 1.091 [0.870 to 1.730] | 0.964 [0.700 to 1.180]
  IFNa : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 4 Post-Vaccination 2 |  | 1.079 [0.780 to 1.480] | 1.252 [0.500 to 1.670]
  IFNa : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNa : Day 8 Post-Vaccination 2 |  | 1.164 [0.930 to 1.520] | 0.906 [0.470 to 1.300]
  IFNb : Day 2 Post-Vaccination 1 | 0.907 [0.700 to 1.170] | 0.929 [0.750 to 1.360] | 0.839 [0.760 to 1.110]
  IFNb : Day 4 Post-Vaccination 1 | 0.941 [0.760 to 1.150] | 1.134 [0.850 to 1.450] | 1.092 [0.760 to 1.270]
  IFNb : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNb : Day 8 Post-Vaccination 1 | 1.000 [0.830 to 1.220] |  |
  IFNb : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 29 Post-Vaccination 1 |  | 0.858 [0.670 to 1.060] | 0.968 [0.880 to 1.260]
  IFNb : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 2 Post-Vaccination 2 |  | 1.172 [1.050 to 1.740] | 0.989 [0.810 to 1.200]
  IFNb : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 4 Post-Vaccination 2 |  | 1.051 [1.000 to 1.200] | 1.033 [0.820 to 1.170]
  IFNb : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNb : Day 8 Post-Vaccination 2 |  | 1.249 [1.000 to 1.530] | 1.074 [0.740 to 1.280]
  IFNy : Day 2 Post-Vaccination 1 | 0.993 [0.940 to 1.160] | 1.118 [1.020 to 1.570] | 0.987 [0.910 to 1.030]
  IFNy : Day 4 Post-Vaccination 1 | 1.049 [0.940 to 1.140] | 1.018 [0.870 to 1.110] | 0.991 [0.930 to 1.020]
  IFNy : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IFNy : Day 8 Post-Vaccination 1 | 1.018 [0.940 to 1.090] |  |
  IFNy : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 29 Post-Vaccination 1 |  | 1.085 [0.930 to 1.190] | 0.958 [0.840 to 1.180]
  IFNy : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 2 Post-Vaccination 2 |  | 1.819 [1.070 to 2.500] | 0.968 [0.930 to 1.030]
  IFNy : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 4 Post-Vaccination 2 |  | 0.854 [0.770 to 0.960] | 0.927 [0.870 to 1.110]
  IFNy : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IFNy : Day 8 Post-Vaccination 2 |  | 0.973 [0.800 to 1.070] | 0.927 [0.850 to 1.010]
  ITAC : Day 2 Post-Vaccination 1 | 0.975 [0.870 to 1.220] | 1.149 [0.980 to 1.290] | 0.926 [0.800 to 1.270]
  ITAC : Day 4 Post-Vaccination 1 | 1.020 [0.860 to 1.360] | 1.160 [0.990 to 1.260] | 0.953 [0.750 to 1.170]
  ITAC : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  ITAC : Day 8 Post-Vaccination 1 | 0.874 [0.610 to 1.460] |  |
  ITAC : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 29 Post-Vaccination 1 |  | 0.895 [0.810 to 1.070] | 0.913 [0.760 to 0.980]
  ITAC : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 2 Post-Vaccination 2 |  | 2.277 [1.350 to 3.660] | 0.916 [0.840 to 0.990]
  ITAC : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 4 Post-Vaccination 2 |  | 1.098 [0.900 to 1.260] | 0.852 [0.660 to 1.210]
  ITAC : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  ITAC : Day 8 Post-Vaccination 2 |  | 1.325 [0.800 to 2.190] | 1.041 [0.910 to 1.210]

9. Secondary Outcome: Fold Change in Cytokine and Chemokine Concentrations From Pre-vaccination - Part 2
Description: Venous blood samples for plasma were used for this assay. A Luminex assay was used to measure concentrations in ng/L. Concentrations for 17 of the total 24 cytokines and chemokines were measured: IL-1b, IL-10, IL-13, IL-2, IL-21, IL-23, IL-4, IL-5, IL-6, IL-7, IL-8, IL-12p70, IL-17A, MIP1a, MIP1b, MIP3a, and TNF-a.
  If no cytokine or chemokine measurements were collected, number of participants is reported as 0.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: fold change
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10 | 10
fold change
  IL-1b : Day 2 Post-Vaccination 1 | 0.981 [0.840 to 1.150] | 0.933 [0.860 to 1.070] | 0.950 [0.880 to 1.160]
  IL-1b : Day 4 Post-Vaccination 1 | 1.050 [0.900 to 1.210] | 1.004 [0.830 to 1.280] | 0.996 [0.800 to 1.120]
  IL-1b : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-1b : Day 8 Post-Vaccination 1 | 0.989 [0.850 to 1.080] |  |
  IL-1b : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 29 Post-Vaccination 1 |  | 1.022 [0.980 to 1.280] | 0.938 [0.800 to 1.120]
  IL-1b : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 2 Post-Vaccination 2 |  | 0.942 [0.810 to 1.340] | 0.940 [0.890 to 1.190]
  IL-1b : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 4 Post-Vaccination 2 |  | 0.890 [0.780 to 1.020] | 1.044 [0.860 to 1.220]
  IL-1b : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-1b : Day 8 Post-Vaccination 2 |  | 1.106 [0.780 to 1.280] | 0.957 [0.810 to 1.070]
  IL-10 : Day 2 Post-Vaccination 1 | 1.106 [0.900 to 1.210] | 1.028 [0.870 to 1.190] | 0.975 [0.840 to 1.120]
  IL-10 : Day 4 Post-Vaccination 1 | 1.043 [0.920 to 1.300] | 1.118 [0.950 to 1.250] | 1.003 [0.810 to 1.160]
  IL-10 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-10 : Day 8 Post-Vaccination 1 | 0.979 [0.810 to 1.120] |  |
  IL-10 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 29 Post-Vaccination 1 |  | 1.076 [0.960 to 1.500] | 1.032 [0.790 to 1.180]
  IL-10 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 2 Post-Vaccination 2 |  | 1.099 [0.910 to 1.290] | 0.919 [0.850 to 0.980]
  IL-10 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 4 Post-Vaccination 2 |  | 0.950 [0.840 to 1.130] | 0.962 [0.770 to 1.150]
  IL-10 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-10 : Day 8 Post-Vaccination 2 |  | 0.979 [0.830 to 1.210] | 0.875 [0.760 to 1.010]
  IL-13 : Day 2 Post-Vaccination 1 | 1.021 [0.940 to 1.090] | 1.024 [0.910 to 1.100] | 0.982 [0.830 to 1.170]
  IL-13 : Day 4 Post-Vaccination 1 | 1.059 [0.970 to 1.180] | 0.988 [0.950 to 1.070] | 0.994 [0.870 to 1.050]
  IL-13 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-13 : Day 8 Post-Vaccination 1 | 1.065 [0.880 to 1.110] |  |
  IL-13 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 29 Post-Vaccination 1 |  | 1.074 [0.840 to 1.420] | 0.990 [0.890 to 1.190]
  IL-13 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 2 Post-Vaccination 2 |  | 0.973 [0.900 to 1.050] | 0.988 [0.910 to 1.030]
  IL-13 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 4 Post-Vaccination 2 |  | 0.979 [0.820 to 1.230] | 0.976 [0.900 to 1.010]
  IL-13 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-13 : Day 8 Post-Vaccination 2 |  | 1.013 [0.770 to 1.130] | 0.975 [0.890 to 1.040]
  IL-2 : Day 2 Post-Vaccination 1 | 1.055 [0.960 to 1.280] | 0.994 [0.960 to 1.030] | 0.964 [0.860 to 1.070]
  IL-2 : Day 4 Post-Vaccination 1 | 1.020 [0.890 to 1.210] | 1.024 [0.910 to 1.240] | 0.908 [0.850 to 1.110]
  IL-2 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-2 : Day 8 Post-Vaccination 1 | 1.080 [0.760 to 1.090] |  |
  IL-2 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 29 Post-Vaccination 1 |  | 1.119 [0.860 to 1.850] | 0.997 [0.710 to 1.140]
  IL-2 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 2 Post-Vaccination 2 |  | 1.059 [0.680 to 1.170] | 0.901 [0.830 to 1.030]
  IL-2 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 4 Post-Vaccination 2 |  | 0.907 [0.690 to 1.090] | 1.023 [0.780 to 1.160]
  IL-2 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-2 : Day 8 Post-Vaccination 2 |  | 1.031 [0.740 to 1.280] | 0.927 [0.840 to 0.970]
  IL-21 : Day 2 Post-Vaccination 1 | 1.152 [0.930 to 1.420] | 0.992 [0.850 to 1.150] | 0.932 [0.850 to 1.210]
  IL-21 : Day 4 Post-Vaccination 1 | 1.402 [0.920 to 1.550] | 0.959 [0.790 to 1.260] | 0.902 [0.840 to 1.070]
  IL-21 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-21 : Day 8 Post-Vaccination 1 | 1.149 [0.750 to 1.330] |  |
  IL-21 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 29 Post-Vaccination 1 |  | 1.213 [1.150 to 1.440] | 0.916 [0.860 to 1.080]
  IL-21 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 2 Post-Vaccination 2 |  | 1.099 [0.950 to 1.280] | 1.040 [0.850 to 1.060]
  IL-21 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 4 Post-Vaccination 2 |  | 0.932 [0.770 to 1.030] | 0.924 [0.790 to 1.210]
  IL-21 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-21 : Day 8 Post-Vaccination 2 |  | 0.861 [0.620 to 1.180] | 0.880 [0.720 to 1.180]
  IL-23 : Day 2 Post-Vaccination 1 | 0.907 [0.820 to 1.060] | 0.998 [0.890 to 1.120] | 0.929 [0.830 to 1.300]
  IL-23 : Day 4 Post-Vaccination 1 | 1.014 [0.780 to 1.470] | 1.006 [0.810 to 1.270] | 0.949 [0.820 to 1.230]
  IL-23 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-23 : Day 8 Post-Vaccination 1 | 0.930 [0.690 to 1.060] |  |
  IL-23 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 29 Post-Vaccination 1 |  | 1.041 [0.910 to 1.280] | 0.993 [0.720 to 1.180]
  IL-23 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 2 Post-Vaccination 2 |  | 1.046 [0.890 to 1.240] | 0.956 [0.880 to 1.190]
  IL-23 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 4 Post-Vaccination 2 |  | 1.032 [0.800 to 1.210] | 0.982 [0.700 to 1.280]
  IL-23 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-23 : Day 8 Post-Vaccination 2 |  | 0.954 [0.770 to 1.460] | 0.979 [0.790 to 1.070]
  IL-4 : Day 2 Post-Vaccination 1 | 0.992 [0.850 to 1.180] | 1.038 [0.930 to 1.130] | 1.034 [0.910 to 1.240]
  IL-4 : Day 4 Post-Vaccination 1 | 1.013 [0.830 to 1.270] | 1.028 [0.840 to 1.170] | 0.921 [0.840 to 1.130]
  IL-4 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-4 : Day 8 Post-Vaccination 1 | 0.969 [0.870 to 1.160] |  |
  IL-4 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 29 Post-Vaccination 1 |  | 1.038 [0.910 to 1.190] | 1.014 [0.870 to 1.170]
  IL-4 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 2 Post-Vaccination 2 |  | 1.014 [0.830 to 1.150] | 0.969 [0.860 to 1.060]
  IL-4 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 4 Post-Vaccination 2 |  | 0.983 [0.830 to 1.130] | 0.935 [0.740 to 1.130]
  IL-4 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-4 : Day 8 Post-Vaccination 2 |  | 1.083 [0.890 to 1.160] | 0.910 [0.730 to 1.080]
  IL-5 : Day 2 Post-Vaccination 1 | 1.062 [0.850 to 1.220] | 1.029 [0.920 to 1.170] | 0.978 [0.840 to 1.100]
  IL-5 : Day 4 Post-Vaccination 1 | 0.986 [0.830 to 1.240] | 1.074 [0.940 to 1.420] | 1.037 [0.770 to 1.270]
  IL-5 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-5 : Day 8 Post-Vaccination 1 | 1.009 [0.800 to 1.110] |  |
  IL-5 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 29 Post-Vaccination 1 |  | 1.010 [0.850 to 1.330] | 1.040 [0.900 to 1.150]
  IL-5 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 2 Post-Vaccination 2 |  | 1.122 [0.980 to 1.380] | 0.980 [0.810 to 1.050]
  IL-5 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 4 Post-Vaccination 2 |  | 1.022 [0.940 to 1.190] | 0.960 [0.870 to 1.190]
  IL-5 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-5 : Day 8 Post-Vaccination 2 |  | 1.123 [0.750 to 1.350] | 0.965 [0.770 to 1.030]
  IL-6 : Day 2 Post-Vaccination 1 | 1.123 [1.000 to 1.590] | 1.601 [1.250 to 2.140] | 0.952 [0.920 to 1.140]
  IL-6 : Day 4 Post-Vaccination 1 | 1.075 [0.900 to 1.550] | 0.990 [0.700 to 1.150] | 0.969 [0.890 to 1.180]
  IL-6 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-6 : Day 8 Post-Vaccination 1 | 0.970 [0.630 to 1.130] |  |
  IL-6 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 29 Post-Vaccination 1 |  | 0.921 [0.700 to 1.500] | 0.996 [0.790 to 1.100]
  IL-6 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 2 Post-Vaccination 2 |  | 1.827 [1.190 to 2.680] | 0.942 [0.870 to 1.110]
  IL-6 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 4 Post-Vaccination 2 |  | 0.907 [0.800 to 1.150] | 1.054 [0.750 to 1.210]
  IL-6 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-6 : Day 8 Post-Vaccination 2 |  | 0.921 [0.610 to 1.140] | 0.961 [0.790 to 1.110]
  IL-7 : Day 2 Post-Vaccination 1 | 1.080 [0.840 to 1.220] | 1.010 [0.900 to 1.220] | 0.982 [0.840 to 1.250]
  IL-7 : Day 4 Post-Vaccination 1 | 0.952 [0.680 to 1.310] | 1.009 [0.880 to 1.270] | 0.934 [0.800 to 1.350]
  IL-7 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-7 : Day 8 Post-Vaccination 1 | 1.000 [0.790 to 1.170] |  |
  IL-7 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 29 Post-Vaccination 1 |  | 0.969 [0.880 to 1.010] | 0.976 [0.760 to 1.150]
  IL-7 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 2 Post-Vaccination 2 |  | 0.953 [0.840 to 1.280] | 0.979 [0.860 to 1.070]
  IL-7 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 4 Post-Vaccination 2 |  | 0.816 [0.710 to 1.130] | 0.966 [0.880 to 1.250]
  IL-7 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-7 : Day 8 Post-Vaccination 2 |  | 1.262 [1.020 to 1.460] | 1.022 [0.780 to 1.110]
  IL-8 : Day 2 Post-Vaccination 1 | 1.111 [0.930 to 1.340] | 1.045 [0.860 to 1.110] | 0.960 [0.890 to 1.070]
  IL-8 : Day 4 Post-Vaccination 1 | 1.073 [0.870 to 1.310] | 0.943 [0.880 to 1.060] | 0.944 [0.810 to 1.070]
  IL-8 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-8 : Day 8 Post-Vaccination 1 | 1.039 [0.900 to 1.070] |  |
  IL-8 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 29 Post-Vaccination 1 |  | 0.970 [0.790 to 1.310] | 0.914 [0.780 to 1.010]
  IL-8 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 2 Post-Vaccination 2 |  | 1.134 [0.940 to 1.280] | 0.988 [0.940 to 1.070]
  IL-8 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 4 Post-Vaccination 2 |  | 0.834 [0.730 to 1.040] | 1.065 [0.890 to 1.180]
  IL-8 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-8 : Day 8 Post-Vaccination 2 |  | 1.299 [0.750 to 1.520] | 0.966 [0.900 to 1.040]
  IL-12p70 : Day 2 Post-Vaccination 1 | 1.048 [0.930 to 1.200] | 1.029 [0.840 to 1.150] | 0.869 [0.730 to 1.100]
  IL-12p70 : Day 4 Post-Vaccination 1 | 1.057 [0.920 to 1.140] | 1.029 [0.940 to 1.260] | 0.916 [0.810 to 1.030]
  IL-12p70 : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-12p70 : Day 8 Post-Vaccination 1 | 1.012 [0.780 to 1.100] |  |
  IL-12p70 : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 29 Post-Vaccination 1 |  | 1.052 [0.950 to 1.600] | 1.059 [0.650 to 1.140]
  IL-12p70 : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 2 Post-Vaccination 2 |  | 1.026 [0.860 to 1.240] | 1.002 [0.810 to 1.150]
  IL-12p70 : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 4 Post-Vaccination 2 |  | 0.933 [0.890 to 1.030] | 1.041 [0.800 to 1.400]
  IL-12p70 : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-12p70 : Day 8 Post-Vaccination 2 |  | 0.901 [0.820 to 1.220] | 0.936 [0.750 to 1.150]
  IL-17A : Day 2 Post-Vaccination 1 | 1.011 [0.950 to 1.160] | 1.074 [0.920 to 1.120] | 0.932 [0.850 to 1.040]
  IL-17A : Day 4 Post-Vaccination 1 | 1.053 [0.860 to 1.200] | 1.019 [0.920 to 1.180] | 0.911 [0.880 to 1.010]
  IL-17A : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  IL-17A : Day 8 Post-Vaccination 1 | 0.965 [0.940 to 1.120] |  |
  IL-17A : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 29 Post-Vaccination 1 |  | 1.153 [1.010 to 1.320] | 0.908 [0.790 to 1.170]
  IL-17A : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 2 Post-Vaccination 2 |  | 0.970 [0.920 to 1.060] | 0.988 [0.910 to 1.020]
  IL-17A : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 4 Post-Vaccination 2 |  | 0.913 [0.820 to 0.980] | 0.999 [0.840 to 1.1170]
  IL-17A : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  IL-17A : Day 8 Post-Vaccination 2 |  | 0.891 [0.610 to 1.170] | 0.956 [0.750 to 1.030]
  MIP1a : Day 2 Post-Vaccination 1 | 1.024 [0.950 to 1.110] | 1.035 [0.990 to 1.040] | 0.963 [0.930 to 1.120]
  MIP1a : Day 4 Post-Vaccination 1 | 1.089 [0.930 to 1.170] | 1.037 [0.940 to 1.110] | 0.997 [0.920 to 1.080]
  MIP1a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP1a : Day 8 Post-Vaccination 1 | 0.966 [0.910 to 1.060] |  |
  MIP1a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 29 Post-Vaccination 1 |  | 1.049 [0.870 to 1.170] | 1.018 [0.850 to 1.080]
  MIP1a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 2 Post-Vaccination 2 |  | 1.018 [0.960 to 1.140] | 1.008 [0.910 to 1.050]
  MIP1a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 4 Post-Vaccination 2 |  | 0.961 [0.850 to 1.060] | 0.978 [0.920 to 1.110]
  MIP1a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1a : Day 8 Post-Vaccination 2 |  | 1.097 [0.960 to 1.230] | 0.970 [0.890 to 1.040]
  MIP1b : Day 2 Post-Vaccination 1 | 1.192 [0.880 to 1.270] | 1.187 [0.940 to 1.330] | 0.955 [0.910 to 1.090]
  MIP1b : Day 4 Post-Vaccination 1 | 1.027 [0.810 to 1.180] | 1.030 [0.990 to 1.200] | 1.023 [0.860 to 1.210]
  MIP1b : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP1b : Day 8 Post-Vaccination 1 | 1.038 [1.010 to 1.070] |  |
  MIP1b : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 29 Post-Vaccination 1 |  | 0.958 [0.810 to 1.190] | 0.942 [0.840 to 1.050]
  MIP1b : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 2 Post-Vaccination 2 |  | 1.576 [1.240 to 2.210] | 0.950 [0.900 to 1.130]
  MIP1b : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 4 Post-Vaccination 2 |  | 0.985 [0.840 to 1.070] | 1.111 [0.850 to 1.220]
  MIP1b : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP1b : Day 8 Post-Vaccination 2 |  | 1.194 [0.860 to 1.320] | 0.960 [0.870 to 1.100]
  MIP3a : Day 2 Post-Vaccination 1 | 1.085 [0.820 to 1.250] | 0.979 [0.820 to 1.010] | 0.968 [0.800 to 1.090]
  MIP3a : Day 4 Post-Vaccination 1 | 1.056 [0.910 to 1.150] | 0.990 [0.820 to 1.130] | 0.976 [0.850 to 1.060]
  MIP3a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  MIP3a : Day 8 Post-Vaccination 1 | 0.976 [0.930 to 1.190] |  |
  MIP3a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 29 Post-Vaccination 1 |  | 0.945 [0.900 to 1.080] | 0.891 [0.720 to 1.110]
  MIP3a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 2 Post-Vaccination 2 |  | 1.033 [0.900 to 1.160] | 0.943 [0.850 to 1.230]
  MIP3a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 4 Post-Vaccination 2 |  | 1.036 [0.910 to 1.200] | 1.021 [0.930 to 1.250]
  MIP3a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  MIP3a : Day 8 Post-Vaccination 2 |  | 1.055 [0.910 to 1.570] | 1.076 [0.900 to 1.670]
  TNF-a : Day 2 Post-Vaccination 1 | 1.022 [1.000 to 1.360] | 1.132 [0.940 to 1.200] | 0.929 [0.850 to 1.080]
  TNF-a : Day 4 Post-Vaccination 1 | 0.965 [0.920 to 1.330] | 1.148 [0.990 to 1.290] | 1.070 [0.860 to 1.180]
  TNF-a : Day 8 Post-Vaccination 1: number analyzed (Participants) | 10 | 0 | 0
  TNF-a : Day 8 Post-Vaccination 1 | 0.998 [0.880 to 1.070] |  |
  TNF-a : Day 29 Post-Vaccination 1: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 29 Post-Vaccination 1 |  | 0.977 [0.820 to 1.240] | 0.869 [0.790 to 1.060]
  TNF-a : Day 2 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 2 Post-Vaccination 2 |  | 1.634 [1.380 to 1.950] | 1.009 [0.880 to 1.180]
  TNF-a : Day 4 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 4 Post-Vaccination 2 |  | 1.112 [0.890 to 1.220] | 1.047 [0.840 to 1.320]
  TNF-a : Day 8 Post-Vaccination 2: number analyzed (Participants) | 0 | 10 | 10
  TNF-a : Day 8 Post-Vaccination 2 |  | 1.199 [0.770 to 1.460] | 0.984 [0.890 to 1.160]

10. Secondary Outcome: Percentage of Participants Achieving Seroconversion Based on Neut Titer (A/H7N9 Vaccine, With and Without Adjuvant)
Description: Seroconversion is defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer =>1:40 or a pre-vaccination Neut titer =>1:10 and a minimum four-fold rise in post-vaccination Neut titer. Venous blood samples for serum were used for this assay. Neut based on the H7N9 strain A/Shanghai/02/2013xPR8 were assessed.
Time Frame: Day 29 Post-Vaccination 2 (Day 57)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10
percentage of participants | 100 [69.2 to 100.0] | 0 [0.0 to 30.8]

11. Secondary Outcome: Percentage of Participants Achieving Seroconversion Based on Neut Titer (A/H3N2v Vaccine)
Description: Seroconversion is defined as either a pre-vaccination Neut titer <1:10 and a post-vaccination Neut titer =>1:40 or a pre-vaccination Neut titer =>1:10 and a minimum four-fold rise in post-vaccination Neut titer. Venous blood samples for serum were used for this assay. Neut based on the H3N2 strain A/Minnesota/11/2010 were assessed.
Time Frame: Day 29 Post-Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A/H3N2v
Number analyzed (Participants) | 10
percentage of participants | 40 [12.2 to 73.8]

12. Secondary Outcome: Geometric Mean Titers of Serum HAI Antibody (A/H7N9 Vaccine, With and Without Adjuvant)
Description: Venous blood samples for serum were used for this assay. HAI based on the H7N9 strain A/Shanghai/02/2013xPR8 were assessed.
Time Frame: Day 1 Pre-Vaccination 1, Day 29 Post-Vaccination 1 (Day 29), and Day 29 Post-Vaccination 2 (Day 57)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10
titer
  Day 1 (Pre-Vaccination 1) | 5.2 [4.8 to 5.6] | 5.0 [NA to NA] — Value is N/A because all subjects had the same value, so no 95% CI is presented.
  Day 29 (Post-Vaccination 1) | 7.3 [4.2 to 12.9] | 5.2 [4.8 to 5.6]
  Day 29 (Post-Vaccination 2) | 85.7 [26.7 to 275.6] | 5.0 [NA to NA] — Value is N/A because all subjects had the same value, so no 95% CI is presented.

13. Secondary Outcome: Geometric Mean Titers of Serum HAI Antibody (A/H3N2v Vaccine)
Description: Venous blood samples for serum were used for this assay. HAI based on the H3N2 strain A/Minnesota/11/2010 were assessed.
Time Frame: Day 1 Pre-Vaccination 1 (Day 1), Day 29 Post-Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | A/H3N2v
Number analyzed (Participants) | 10
titer
  Day 1 Pre-Vaccination 1 | 37.3 [16.4 to 85.1]
  Day 29 Post-Vaccination 1 | 144.2 [44.8 to 464.2]

14. Secondary Outcome: Geometric Mean Titers of Serum Neut Antibody (A/H7N9 Vaccine, With and Without Adjuvant)
Description: Venous blood samples for serum were used for this assay. Neut based on the H7N9 strain A/Shanghai/02/2013xPR8 were assessed.
Time Frame: Day 1 Pre-Vaccination 1 (Day 1), Day 29 Post-Vaccination 1 (Day 29), and Day 29 Post-Vaccination 2 (Day 57)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | A/H7N9 + AS03 | A/H7N9
Number analyzed (Participants) | 10 | 10
titer
  Day 1 (Pre-Vaccination 1) | 5.0 [NA to NA] — Value is N/A because all subjects had the same value, so no 95% CI is presented. | 5.0 [NA to NA] — Value is N/A because all subjects had the same value, so no 95% CI is presented.
  Day 29 (Post-Vaccination 1) | 17.4 [11.6 to 26.2] | 5.4 [4.6 to 6.3]
  Day 29 (Post-Vaccination 2) | 190.3 [112.5 to 321.9] | 5.9 [4.5 to 7.8]

15. Secondary Outcome: Geometric Mean Titers of Serum Neut Antibody (A/H3N2v Vaccine)
Description: Venous blood samples for serum were used for this assay. Neut based on the H3N2 strain A/Minnesota/11/2010 were assessed.
Time Frame: Day 1 Pre-Vaccination 1 (Day 1), Day 29 Post-Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | A/H3N2v
Number analyzed (Participants) | 10
titer
  Day 1 Pre-Vaccination 1 | 171.5 [86.1 to 341.7]
  Day 29 Post-Vaccination 1 | 485.0 [229.9 to 1023.2]

ADVERSE EVENTS:
Time Frame: For all arms, solicited Adverse Events (AEs) were collected from the time of each study vaccination through 8 days post-vaccination and unsolicited AEs were collected from the time of first study vaccination through 28 days after last study vaccination. For the A/H7N9 and A/H7N9 + AS03 arms, Serious Adverse Events (SAEs) and Medically Attended Adverse Events (MAAEs) were additionally collected from the time of first study vaccination through 12 months after last study vaccination.
Description: Solicited AEs include injection site reactions and systemic reactions. Injection site reactions include pruritus, ecchymosis, erythema, induration/swelling, pain, and tenderness. Systemic reactions include fever, feverishness, fatigue, malaise, myalgia (exclusive of the injection site), arthralgia (exclusive of the injection site), headache, and nausea.
Groups:
- A/H3N2v: One dose of 15 ug of A/H3N2v virus vaccine at Day 1
- A/H7N9 + AS03: Two doses of 3.75 µg of AH7N9 virus vaccine + AS03 adjuvant at Day 1 and Day 29
- A/H7N9 + PBS: Two doses of 3.75 µg of A/H7N9 virus vaccine at Day 1 and Day 29
Arm/Group | A/H3N2v | A/H7N9 + AS03 | A/H7N9 + PBS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 8/10 | 10/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/H3N2v (N=10) | A/H7N9 + AS03 (N=10) | A/H7N9 + PBS (N=10)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/H3N2v (N=10) | A/H7N9 + AS03 (N=10) | A/H7N9 + PBS (N=10)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Fatigue (General disorders) | 2 (2) | 7 (10) | 3 (3)
Feeling Hot (General disorders) | 0 (0) | 4 (4) | 3 (3)
Injection Site Erythema (General disorders) | 2 (2) | 7 (10) | 1 (1)
Injection Site Haemorrhage (General disorders) | 0 (0) | 3 (3) | 0 (0)
Injection Site Induration (General disorders) | 0 (0) | 3 (3) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 8 (12) | 0 (0)
Injection Site Pain (Tenderness) (General disorders) | 6 (6) | 10 (18) | 2 (2)
Malaise (General disorders) | 1 (1) | 6 (6) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT02921997/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT02921997/SAP_001.pdf